CLINICAL TRIAL: NCT00438867
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Ad5FGF-4 in Female Patients With Stable Angina Pectoris Who Are Not Candidates for Revascularization
Brief Title: Angiogenesis in Women With Angina Pectoris Who Are Not Candidates for Revascularization
Acronym: AWARE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardium Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-3-001
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2008-11

CONDITIONS: Angina Pectoris
Keywords: angina; FGF-4; angiogenesis; growth factor; myocardia ischemia; revascularization
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Genetic: Ad5FGF-4
- 2 (Experimental)
  Interventions: Genetic: Ad5FGF-4
- 3 (Placebo Comparator)
  Interventions: Genetic: Placebo

INTERVENTIONS:
Genetic: Ad5FGF-4 — Adenovirus serotype-5 mediated human fibroblast growth factor-4 gene transfer
  Arms: 1; 2
Genetic: Placebo — Control group
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether a one-time intracoronary infusion of Ad5FGF-4 is effective in reducing the time to onset myocardial ischemia as measured by exercise treadmill testing and improving myocardial blood flow as measured by SPECT imaging. Exercise capacity, angina functional class, patient symptoms and quality of life will also be evaluated to characterize the efficacy of Ad5FGF-4. Short-term and long-term safety of Ad5FGF-4 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18-75 years of age inclusive
* Stable angina classified as CCS III or IV
* Receiving treatment with at least two classes of chronic anti-anginal medication, of which two are at the maximally tolerated dose
* Left ventricular ejection fraction (LVEF) of ≥30%
* Not a candidate for, or unlikely to benefit from standard revascularization procedures as verified by an independent cardiologist or cardiothoracic surgeon (not a study investigator) at each center
* Can undergo ETT using the modified Bruce protocol and;

  1. ECG changes diagnostic of myocardial ischemia occur during the first 10 minutes of exercise
  2. Variability of the time to onset of ECG changes diagnostic of myocardial ischemia is ≤25% or within 60 seconds if the time to onset of myocardial ischemia occurs within the first 4 minutes of exercise as determined by two consecutive screening treadmill tests
* Evidence of stress induced myocardial ischemia by adenosine SPECT, defined as a reversible perfusion defect size of ≥9%
* Willing and able to comply with the study requirements including long-term follow-up
* Provided written informed consent

Exclusion Criteria:

* Patients of childbearing potential (must be surgically sterile or post-menopausal)
* Patients for whom an immediate revascularization procedure is indicated (CABG surgery or PCI)
* Myocardial infarction within the past 3 months
* Unstable angina or hospitalization requiring intravenous anti-anginal therapy within the 14 days prior to the start of screening evaluations
* Congestive heart failure NYHA Class IV
* Electrocardiogram that precludes accurate assessment of exercise induced myocardial ischemia (e.g., left bundle branch block, Wolf-Parkinson-White syndrome, atrial fibrillation)
* Myocarditis or restrictive pericarditis
* Left main coronary stenosis ≥70% (unless the patient has a patent graft or collateral vessels supplying the left coronary circulation) or proximal stenoses ≥70% in all major coronary conduit vessels (coronary arteries and bypass grafts)
* Clinically significant aortic or mitral valvular heart disease
* Coronary ostial stenosis that precludes adequate catheter engagement in any target vessel
* Coronary artery to venous communications, which bypass the coronary capillary bed
* Untreated life-threatening ventricular arrhythmias
* CABG surgery within the past 6 months, unless those grafts are now occluded.
* Percutaneous transluminal angioplasty (PTCA) within the past 3 months, unless the dilated vessel(s) are now occluded
* Enhanced external counterpulsation (EECP) within 3 months prior to the start of screening evaluations
* Transmyocardial or percutaneous myocardial laser revascularization within the previous year
* Prior treatment with any cardiovascular gene or stem cell therapy.
* Any intercurrent illness that may interfere with their ability to perform a maximal ETT
* Any major organ disease that substantially impairs life expectancy.
* History of cancer, other than basal cell carcinoma, or patients with any laboratory or physical exam or diagnostic procedure finding suggestive of current malignancy
* Moderate to severe nonproliferative or proliferative retinopathy from any cause (ETDRS score >35), clinically significant macular edema, or previous panretinal photocoagulation therapy
* Heparin induced thrombocytopenia or history of idiopathic thrombocytopenic purpura or other medical condition causing thrombocytopenia
* SGPT level greater than 2.0 times the upper limit of the laboratory normal range
* Bilirubin level ≥2.0 mg/dL
* Serum creatinine ≥2.5 mg/dL
* Platelet count <100,000/μL
* White blood cell count <3,000/μL
* Positive test for hepatitis B or C
* Positive test for HIV
* History of colon cancer in a first degree relative (i.e., parent, sibling or offspring) unless the patient has undergone a colonoscopy in the past 36 months with negative findings
* History of breast cancer in a first degree relative
* Patient in a family with any documented hereditary cancer syndrome
* Prior anaphylaxis reaction to iodinated contrast agents
* Patients who are known to be immunosuppressed or are receiving chronic treatment with immunosuppressive drugs
* Received an investigational drug or biologic within 30 days of screening or are currently participating in an investigational drug, biologic or device trial

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in time to onset of ECG changes diagnostic of myocardial ischemia during ETT | Month 6

SECONDARY OUTCOMES:
Change in reversible perfusion defect size as measured by adenosine single-photon emission computed tomography with technetium-99m sestamibi (SPECT)(principal secondary endpoint) | Month 6
Change in total exercise treadmill time | Months 3, 6 and 12
Change in time to onset ECG changes diagnostic myocardial ischemia during ETT | Months 3 and 12
Change in time to onset of angina during ETT | Months 3, 6 and 12
Change in angina frequency and nitroglycerin | Months 3 and 6
Change in patient functional status using CCS angina class | Months 3, 6 and 12
Change in rest and stress left ventricular ejection fraction assessed using gated SPECT | Month 6
Change in quality of life using the Seattle Angina Questionnaire | Months 6 and 12
Safety of Ad5FGF-4 as assessed by adverse events and clinical laboratory testing | Through month 12
Long-term safety of Ad5FGF-4 as assessed by clinically important events | Through month 60

CONTACTS AND LOCATIONS:
Overall Officials: Robert Engler, MD, Study Director — Cardium Therapeutics
Locations (47):
- United States (47):
  - University of Alabama, Birmingham, Alabama
  - Banner Heart Hospital, Phoenix, Arizona
  - Southwest Heart, Tucson, Arizona
  - Access Clinical Trials, Beverly Hills, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mission Internal Medical Group, Mission Viejo, California
  - UCSD Medical Center, San Diego, California
  - Aurora Denver Cardiology, Aurora, Colorado
  - South Denver Cardiology, Littleton, Colorado
  - Cardiovascular Research Institute, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Florida Hospital, Orlando, Florida
  - St Joseph's Research Institute, Atlanta, Georgia
  - St. Luke's Idaho Cardiology Associates, Boise, Idaho
  - Fox Valley Cardiovascular Consultants, Aurora, Illinois
  - Midwest Heart Foundation, Lombard, Illinois
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - The Care Group, Indianapolis, Indiana
  - Cardiovascular Associates, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Duluth Clinic, Duluth, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mid America Heart Institute, Kansas City, Missouri
  - St. Anthony's Medical Center, St Louis, Missouri
  - BryanLGH Heart Institute, Lincoln, Nebraska
  - Creighton University, Omaha, Nebraska
  - The Valley Hospital, Ridgewood, New Jersey
  - Lenox Hill Heart & Vascular Institute, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - North Ohio Heart Center, Elyria, Ohio
  - Oklahoma Cardiovascular Associates, Oklahoma City, Oklahoma
  - Providence Heart & Vascular Institute, Portland, Oregon
  - Heritage Cardiology Associates, Camp Hill, Pennsylvania
  - Geisinger Clinic, Danville, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - The Stern Cardiovascular Center, Germantown, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Baylor University Medical Center at Dallas, Dallas, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Swedish Medical Center, Seattle, Washington
  - Care Foundation, Wausau, Wisconsin

REFERENCES:
- [Derived] Henry TD, Grines CL, Watkins MW, Dib N, Barbeau G, Moreadith R, Andrasfay T, Engler RL. Effects of Ad5FGF-4 in patients with angina: an analysis of pooled data from the AGENT-3 and AGENT-4 trials. J Am Coll Cardiol. 2007 Sep 11;50(11):1038-46. doi: 10.1016/j.jacc.2007.06.010. Epub 2007 Aug 24. PMID 17825712